CLINICAL TRIAL: NCT06425289
Title: Macrohemodynamic Impact of Fluid Removal With Net Ultrafiltration in Patients With Continuous Renal Replacement Therapy: A Monocentric Ancillary Study of the EarlyDry Randomized Controlled Trial
Brief Title: Macrohemodynamic Impact of Fluid Removal With Net Ultrafiltration in Patients With Continuous Renal Replacement Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_5388
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Fluid Removal; Critically Ill; Continuous Renal Replacement Therapy; Fluid Overload
Keywords: Fluid removal; Hemodynamic; Net ultrafiltration; Continuous renal replacement therapy
MeSH Terms: conditions — Critical Illness; Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Corrective strategy: Procedure: Fluid balance negativation
  During the RRT, UFnet will be settled on 2ml/kg/h and adapted to hemodynamic tolerance and tissue perfusion .
  When the patient's baseline body weight is reached the UF net will be settled to maintain it.
  In case of failure of the fluid balance negativation after 24h, UFnet will be settled on 3ml/kg/h. Then when the baseline body weight is reached UFnet will be settled on 0.5 et 1ml/kg/h or if necessary adapted to 1,5ml/kg/h to maintain it
  In case of hemodynamic intolerance (NADN > 0,5 µg/kg/min) or tissue hypoperfusion, UF net will be stopped during 6 hours and restarted if NADN < 0,5 µg/kg/min and without tissue hypoperfusion.
  Interventions: Other: Macrohemodynamic parameters
- Other: Stabilizing strategy In the control group, all patients will have a UFnet 2 ml settled: Procedure: Body weight Stabilization
  During the RRT, UFnet will be settled between 0 et 1 ml/kg/h and adapted in case of weight stabilization failure or hemodynamic intolerance.
  In case of weight stabilisation failure (variation >5%), the UF net can be increased to 1,5 ml/kg/h.
  In case of hemodynamic intolerance (NADN > 0,5 µg/kg/min), UF net will be stopped during 6 hours and restarted if NADN < 0,5 µg/kg/min.
  Interventions: Other: Macrohemodynamic parameters

INTERVENTIONS:
Other: Macrohemodynamic parameters — Macrohemodynamic parameters will be estimated with transpulmonary thermodilution every 6 hours during the intervention period (5 days).
  * Cardiac index
  * Extravascular lung water index
  * Pulmonary vascular permeability index
  * Cardiac function index
  * Global end-diastolic volume index
  * Central venous pressure
  * Fluid responsivness status (passive leg rising test)

SUMMARY:
Macrohemodynamic impact of fluid removal with net ultrafiltration in patients with continuous renal replacement therapy. A monocentric ancillary study of the EarlyDry randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute kidney injury treated by continuous renal replacement therapy in ICU less than 7 days,
* At least 1 organ failure during ICU in addition to AKI (mechanical ventilation or vasopressors administration>12 hours),
* Cumulative UF net less than 1000ml before inclusion,
* Norepinephrine < 0,5 µg/kg/min,
* Absence of hypoperfusion signs,
* Fluid overload defined as follows: fluid overload > 5% of base weight (based on cumulative fluid balance or a weight gain) and/or peripheral edema (AKIKI edema scale > 2).

Exclusion Criteria:

* Chronic renal failure hemodialyzed before admission to the ICU,
* Mechanical circulatory support (ECMO, LVAD),
* Pregnant, child -bearing age or lactating women,
* Stroke less than 30 days,
* Intestinal ischemia less than 7 days documented non-operated,
* Interventional study participation or exclusion period on going,
* Guardianship, curatorship or safeguard of justice,
* Absence of signature of free and informed consent by the patient and/or relative,
* Patients not affiliated to a social security scheme or beneficiaries of a similar scheme
* Absence of transpulmonary thermodilution monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with fluid overload and renal replacement therapy for fluid overload, included in EarlyDry trial (NCT05817539) and monitored with transpulmonary thermodilution.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of a low cardiac index | Every 6 hours between day 0 to day 5 (intervention period)
  Area under the curve of a cardiac index < 2.4 L/min/m2 (L/min/m2.hr), determined by transpulmonary thermodilution every 6 hours, with three boli of cold saline in the superior vena cava territory.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'anesthésie-réanimation, Hôpital Louis Pradel, Hospices Civils de Lyon, Bron, France